CLINICAL TRIAL: NCT05458791
Title: Application of Intra-arterial CT Perfusion During Interventional Radiology
Brief Title: Intra-arterial Perfusion in Interventional Radiology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Other Study IDs: SHA0010
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Computed Tomography; Arterial Perfusion; Liver; Interventional Radiology
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Standard Dose Intra-arterial Perfusion: All patients will undergo standard of care interventional treatment for liver cancer. The procedure will take place utilizing fluoroscopic and CT guidance. During their procedure, patients will have intra-arterial CT perfusion maps derived of the liver including the region of the tumor. (n=10)
  Interventions: Device: Intra-arterial Perfusion
- Low Dose Intra-arterial Perfusion: Investigate the impacts on contrast and radiation doses and the robustness of reconstruction algorithms on intra-arterial CT perfusion using a lower radiation dose technique. (N=10)
  Interventions: Device: Intra-arterial Perfusion

INTERVENTIONS:
Device: Intra-arterial Perfusion — All patients will undergo standard of care locoregional intra-arterial (IA) treatment for HCC. The procedure will take place utilizing fluoroscopic and CT guidance. Following catheterization of the femoral or radial artery, CT angiography of the hepatic circulation will be performed to define the hepatic vascular anatomy. Intra-arterial CT perfusion will be performed prior to IA treatment by the interventional radiologist to understand the dynamics of hepatic circulation or to manage the IA treatment strategy.

SUMMARY:
Patients are being asked to participate in a study to better determine blood flow going to tumors in the liver. They will undergo an embolization procedure in interventional radiology where the goal is to provide treatment directly into the liver tumor. These treatments are delivered into the blood vessels feeding the tumors. Improving these treatments relies on better understanding the blood flow into the tumor. By understanding how much blood flows into the tumors, the goal is to make sure there is the best chance of killing the tumor. The investigators are attempting to use a special type of CT scan during the procedure to determine the blood flow to the tumors.

DETAILED DESCRIPTION:
Accurate liver imaging is critically important for the appropriate management of hepatocellular carcinoma (HCC) patients. The unique capability of the 4 dimensional (4D) CT system that combines CT and vascular imaging in real time has the great potential to provide physiologic and functional information to the operators to help guide therapy decisions during interventional procedures. However, the workflow, protocols and parameters have not been studied and optimized to support the use of perfusion techniques during interventional procedures. Efforts to reduce contrast and radiation doses associated with perfusion imaging to as low as reasonably achievable (ALARA) are also important steps to ensure patient safety while generating clinically meaningful images. Reducing radiation doses may be achieved by adjusting scan parameters, then applying reconstruction techniques to improve the image quality. The new generation of reconstruction algorithms, such as Model-Based iterative reconstruction, or deep-learning reconstruction algorithms (e.g. AiCE), simultaneously improve noise (lower dose) and enhances low contrast characteristics (less contrast). This pilot study aims to demonstrate the use of 4D CT system to acquire liver perfusion information to support the interventional procedure, and to derive as low as reasonably achievable (ALARA) dose levels and examine the robustness of reconstruction algorithms that generate clinically meaningful perfusion maps.

The study will investigate the impact of different dose levels, and the robustness of reconstruction algorithms on CT perfusion maps. A successful study could allow for dissemination of these methods for use to the wider physician audience with an optimum ALARA dose levels. Furthermore, the potential knowledge gained from this study will further educate the medical community about the potential benefits of 4D CT intra-arterial CT perfusion as an adjunct imaging technique and may steer the direction for future larger scale trials and studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 years
2. primary or secondary liver tumor(s)
3. Trans-arterial chemoembolization (TACE) or trans-catheter radio embolization (TARE) approved by multidisciplinary tumor board
4. Tumor in an area without prior surgical or ablative therapy
5. At least 1 tumor greater than 1.5 cm in greatest diameter

   Exclusion Criteria:
6. Not eligible for TACE procedure.
7. Same additional exclusion criteria as aim 1
8. Any residual ethiodized oil accumulation in the liver
9. No prior IA treatment in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 20 patients with primary or secondary liver tumor(s) who undergo TACE intervention will be assigned to one of each group
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of Parameters for Intra-arterial Perfusion | 1 Day to 1 year
  Intra-arterial CT perfusion will be performed prior to IA treatment by the interventional radiologist to understand the dynamics of hepatic circulation or to manage the IA treatment strategy.

SECONDARY OUTCOMES:
Impact of low dose radiation technique on intra-arterial perfusion parameters | 1 Day to 1 Year
  Evaluating low dose radiation on perfusion parameters

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh P Shah, MD, Principal Investigator — VA Palo Alto Health Care System - Interventional Radiology
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moawad AW, Szklaruk J, Lall C, Blair KJ, Kaseb AO, Kamath A, Rohren SA, Elsayes KM. Angiogenesis in Hepatocellular Carcinoma; Pathophysiology, Targeted Therapy, and Role of Imaging. J Hepatocell Carcinoma. 2020 Apr 23;7:77-89. doi: 10.2147/JHC.S224471. eCollection 2020. PMID 32426302